CLINICAL TRIAL: NCT04672772
Title: Retrospective Study With Cetuximab Plus Paclitaxel as First Line for Recurrent and/or Metastatic SCCHN (Squamous Cell Carcinoma of the Head and Neck): Real World Data.
Brief Title: Cetuximab Plus Paclitaxel as First Line for Recurrent and/or Metastatic SCCHN: Real World Data.
Status: Completed | Type: Observational
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: TTCC-2019-02; TTC-CET-2020-01 (Other: Agencia Española del Medicamento y Productos Sanitarios)
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Cetuximab; Paclitaxel; recurrent and/or metastatic; retrospective observational study; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Paclitaxel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recurrent and/or metastatic SCCHN: Patients who received at least one dose of both paclitaxel 80 mg/m2 as a starting dose with weekly cetuximab, that could have been switched to biweekly during the maintenance phase, as a first line regimen in recurrent and/or metastatic disease.
  Interventions: Drug: Cetuximab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cetuximab — Weekly cetuximab at starting dose, that could be switched to biweekly
Drug: Paclitaxel — Paclitaxel at starting dose of 80 mg/m2

SUMMARY:
Retrospective observational study that aims to collect real world data on the cetuximab plus paclitaxel regimen as first line treatment for recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN).

Assignment of a patient to a specific therapeutic strategy has been already decided in the past according to normal routine clinical practice; the decision to prescribe a specific treatment (between January 2012 and December 2018) was clearly dissociated from the decision to include a patient in the present study.

The investigators will retrospectively collect the information for 500 patients diagnosed with recurrent and/or metastatic SCCHN treated with a cetuximab plus paclitaxel regimen as first line for unresectable recurrent and/or metastatic disease, starting treatment with the defined cetuximab plus paclitaxel regimen, in 20 hospital members of the "Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (TTCC)", who express consent to participate in the study or have not explicitly withheld consent for use of their data. The information from the patients' medical records will be collected through the online database of the TTCC Group.

DETAILED DESCRIPTION:
Retrospective observational study that aims to collect real world data on the cetuximab plus paclitaxel regimen as first line treatment for recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN) with the restriction that the data collection will only be clinical data from patients who received paclitaxel 80 mg/m2 as a starting dose with weekly cetuximab that could have been switched to biweekly during the maintenance phase.

The main objective will be to estimate the Progression-free survival (PFS) in patients treated with paclitaxel 80 mg/m2 as a starting dose, with weekly cetuximab that could have been switched to biweekly during the maintenance phase, as first line for recurrent and/or metastatic SCCHN.

Secondary objectives include:

To determine the Overall Response Rate (ORR), Best Overall Response (BOR), Disease Control Rate (DCR), overall survival (OS), duration of response (DoR), and safety in patients treated with the defined cetuximab plus paclitaxel regimen.

To evaluate the percentage of long disease-free survivors (defined as patients disease-free and alive at 2 years), and evaluate the percentage of long non-disease-free survivors (defined as patients not disease free, but alive at 2 years.

Analyses of patient outcomes by prognostic subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed recurrent and/or metastatic head and neck squamous-cell carcinoma including oral cavity, oropharynx, hypopharynx and larynx.

Note: Histological confirmation is required at the diagnosis of the primary. Not for recurrence and/or metastatic stages when radiological or clinical confirmation is valid

* Patients who received at least one dose of both paclitaxel 80 mg/m2 as a starting dose with weekly cetuximab, that could have been switched to biweekly during the maintenance phase, as a first line regimen in recurrent and/or metastatic disease.
* Start of first cycle of paclitaxel plus cetuximab between 1 January 2012, and 31 December 2018.
* Aged ≥ 18 years at the time of diagnosis of R/M SCCHN.
* Voluntary written consent, if applicable*

  * Note: Waiver of consent could be acceptable after all reasonable efforts and procedures have been followed and exhausted, and when an explicit refusal to sign the informed consent or refusal for use of data, or a revocation of consent by the patient has not been obtained.

Exclusion Criteria:

* Patients with histologically confirmed R/M SCCHN, who have also an unknown primary tumor or nasopharyngeal cancer or a non-squamous head & neck cancer.
* Patients who received the paclitaxel and cetuximab regimen for the first time in recurrent and/or metastatic disease as a second or subsequent line.
* Eastern Cooperative. Oncology Group (ECOG) performance status > 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with recurrent and/or metastatic SCCHN treated with a cetuximab plus paclitaxel regimen as first line for unresectable R/M disease, starting treatment with the defined cetuximab plus paclitaxel regimen, between January 2012 and December 2018 in 20 hospital members of the "Grupo Español de Tratamiento de Tumores de Cabeza y Cuello", who express consent to participate in the study or have not explicitly withheld consent for use of their data.
Sampling Method: Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, average 1 year
  The PFS time is defined as the time from start of study treatment (first administration of cetuximab or paclitaxel) to the date of progression or death, whichever occurs first. In patients without a PFS event, the PFS time will be censored on the date of the last radiological evaluation or on the date of the last study treatment received if the tumor response has not been evaluated after start of study treatment. If no PFS was observed prior to start of second line treatment, then the PFS time will be censored at the first date of second line treatment.

SECONDARY OUTCOMES:
Best Overall Response (BOR) | Through study completion, average 1 year
  Best overall response during study treatment with the categories complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) or not available (NA), as assessed by the responsible physician. The method used to assess BOR (e.g. RECIST and version) will be also recorded.
Overall Response Rate (ORR) | Through study completion, average 1 year
  Overall response rate, defined as the proportion of patients with CR or PR as BOR.
Disease Control Rate (DCR) | Through study completion, average 1 year
  The proportion of patients with CR, PR or SD as BOR.
Frequency of Adverse Events (AEs) | Through study completion, average 1 year
  Safety will be studied as function of AEs frequency: The number of adverse events classified by type and intensity
Overall survival (OS) | Through study completion, average 1 year
  Defined as time from start of study treatment until date of death due to any cause. In patients without death the OS time is censored at the last date known to be alive.
Relative dose intensity (RDI) | Through study completion, average 1 year
  Relative dose intensity (RDI) defined as amount of drug administered per unit of time expressed as the fraction of that defined in the standard regimen
Dose-related and compliance data | Through study completion, average 1 year
  Frequency and magnitude of dose interruptions, dose modifications and discontinuation of treatment classified by the cause of discontinuation including adverse events, relapse, medical decision, patient decision, death and loss of follow-up.
Duration of Response (DOR) | Through study completion, average 1 year
  Defined as the time from the first occurrence of PR or CR as BOR until PD or death, whichever occurs first in patients with CR or PR as BOR.
  The censoring rules specified for PFS will be also applied for duration of response.
Proportion of long disease-free survivors | Through study completion, average 1 year
  The proportion of patients alive and disease-free at 2 years after start of study treatment. Only disease-free patients under first line treatment should be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Cirauqui Cirauqui, M.D. Ph.D., Principal Investigator — Institut Catalá d'Oncologia (ICO) Badalona; Jordi Rubió Casadevall, M.D. Ph.D., Principal Investigator — Institut Catalá d'Oncologia (ICO) Girona
Locations (20):
- Spain (20):
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Regional Universitario de Málaga, Málaga, Andalusia
  - Hospital Universitario Virgen de Valme, Seville, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Virgen de la Salud, Toledo, Castille-La Mancha
  - Institut Catalá d'Oncologia (ICO) Badalona, Badalona, Catalonia
  - Institut Catalá d'Oncologia (ICO) Girona, Girona, Catalonia
  - Hospital Duran i Reynalds (ICO-Hospitalet), L'Hospitalet de Llobregat, Catalonia
  - Centro Oncológico de Galicia, A Coruña, Galicia
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Complejo Hospitalario Navarra (PAMPLONA), Pamplona, Navarre
  - Hospital Universitario Canarias (TENERIFE), San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital de Mar, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No